CLINICAL TRIAL: NCT05931588
Title: Effect of Pilates Exercises on Postpartum Fatigue, Maternal Functioning and Quality of Life
Brief Title: Pilates Exercises on Postpartum Fatigue, Maternal Functioning and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01366 Ayesha
Record Dates: First submitted 2023-01-04; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Maternal Fatigue
Keywords: Pilates; maternal fatigue; maternal functioning
MeSH Terms: interventions — Respiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercises, streching and breathing (Experimental): the intervention Pilates exercises, streching and breathing exercises is administered under supervision
  Interventions: Other: Pilates excercises, streching and breathing; Other: stretching and breathing
- streching and breathing (Experimental): home based exercise program which is streching and breathing.
  Interventions: Other: stretching and breathing

INTERVENTIONS:
Other: Pilates excercises, streching and breathing — international group receive Pilates exercises, stretching and breathing two times a week (30 min per session) perform 3 to 5 reps of Pilates exercises under supervision
  Arms: Pilates exercises, streching and breathing
Other: stretching and breathing — control group guided with stretching and breathing home based program both group till 8 week both groups

SUMMARY:
The aim of the study is to determine the effect of Pilates exercises on postpartum fatigue, maternal functioning and quality of life.

DETAILED DESCRIPTION:
the effect of Pilates exercises in reducing postpartum fatigue is not well known however in recent study Pilates exercises alone was quantified which was based on home exercises and had a positive effect, it was conducted in primiparas women, there was also possibility of recall bias due to self report nature of data

ELIGIBILITY:
Inclusion Criteria:

* Multiparous females
* Age 18 to 45 years
* Females with vaginal delivery
* Two weeks after Spontaneous Vaginal Delivery
* Fatigue score of >11 on Fatigue Assessment scale

Exclusion Criteria:

* Postpartum depression score greater or equal to 10 , based on the Edinburgh Postnatal Depression scale (EPDS)
* Postpartum anemia
* Generalized Anxiety Disorders
* Chronic illnesses (Diabetes /hypothyroidism)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
postnatal maternal fatigue | 8 Week
  The Postnatal Accumulated Fatigue Scale (PAFS) (Tsuchiya et al., 2016) was once used to investigate maternal fatigue and included questions masking the three areas of physical, emotional and cognitive fatigue. The PAFS involves thirteen objects with every coded on a three-point response ranking the place zero = rarely, 1 = sometimes and three = often. Total rankings vary from zero to 39 with greater ratings indicating a greater stage of fatigue. The PAFS consists of questions overlaying three areas of physical, emotional, and cognitive fatigue and has top validity and interior consistency.

SECONDARY OUTCOMES:
barkin indexmaternal functioning | 8 Week
  The BIMF used to be developed as a multidimensional instrument for measuring maternal functioning in each medical and research settings. It used to be designed in 2010 by way of Barkin et al. This instrument consists of 20 gadgets that cover all factors of maternal functioning, such as self-care, child care, mother-child interaction, household management, psychological well-being, adjustment, and social help.
postnatal quality of life | 8 Week
  The Maternal Postpartum Quality of Life (MAPP-QOL) instrument consisted of 41 items. The instrument was intended to be completed by mothers during the early postpartum period following hospital discharge. The development of the instrument had two parts (satisfaction and importance) Part 1 queried the participant about her satisfaction with each item (1-6), with 1 = very dissatisfied and 6 =very satisfied. Part 2 queried about her level of importance with each item, 1 = very dissatisfied and 6 = very satisfied. Scores reflect individual values as well as satisfaction, producing a more accurate reflection of QOL.

OTHER OUTCOMES:
generalized anxiety scale | 8 Week
  The 7-item Generalized Anxiety Disorders Scale (GAD-7; Spitzer) used to be developed as a screener for generalized anxiousness disease (GAD). The seven objects examine (1) feeling nervous, anxious, or on edge; (2) being in a position to quit or manipulate worrying; (3) stressful tool a whole lot about extraordinary things; (4) bother relaxing; (5) being restless; (6) turning into effortlessly aggravated or irritable; and (7) feeling afraid as if something awful may happen.
• Edinburgh postnatal depression scale (EPDS) | 8 Week
  The EPDS was once delivered in 1987. When at first conceived, this 10-item self-report questionnaire was once designed for use in women in the postnatal period, for the purposes of clinical practice and research.

CONTACTS AND LOCATIONS:
Overall Officials: Summra Andleeb, MS(OMPT), Principal Investigator — riphah internation university
Locations (1):
- Imrana nasir family clinic, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No